CLINICAL TRIAL: NCT04009057
Title: Multi-center, Israeli, Non-interventional, Cohort Study of the Effectiveness, Safety, Adherence, and Health-related Quality of Life in HIV-1 Infected Adult Patients Receiving Bictegravir/ Emtricitabine/Tenofovir Alafenamide (B/F/TAF)
Brief Title: Effectiveness, Safety, Adherence, and Health-related Quality of Life in HIV-1 Infected Adults Receiving Bictegravir/ Emtricitabine/Tenofovir Alafenamide (B/F/TAF)
Acronym: BIC-STaR
Status: Completed | Type: Observational
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Other Study IDs: GS-IL-380-5335
Record Dates: First submitted 2019-07-02; First posted 2019-07-05 (Actual); Last update posted 2022-05-03 (Actual); Status verified 2022-04

CONDITIONS: HIV-1-infection
MeSH Terms: interventions — bictegravir, emtricitabine, tenofovir alafenamide, drug combination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- B/F/TAF: HIV-1 infected adults who initiate B/F/TAF therapy
  Interventions: Other: B/F/TAF

INTERVENTIONS:
Other: B/F/TAF — B/F/TAF administered in accordance with the approved product monograph
  Other Names: Biktarvy®

SUMMARY:
The primary objective of this study is to evaluate HIV-1 RNA suppression, defined as HIV-1 RNA < 50 copies/mL, at 12 months after initiating or switching to bictegravir/ emtricitabine/tenofovir alafenamide (B/F/TAF).

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infection
* Signed informed consent
* Initiating treatment with B/F/TAF

Exclusion Criteria:

* Participation in any interventional clinical trial

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population will be comprised of antiretroviral therapy (ART)-naïve and ART-experienced HIV-1 infected adults aged ≥ 18 years initiating treatment with B/F/TAF in routine clinical care in Israel.
Sampling Method: Non-Probability Sample
Enrollment: 143 (Actual)
Dates: Start 2019-07-09 (Actual); Primary Completion 2022-03-21 (Actual); Study Completion 2022-03-21 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants with HIV-1 RNA Suppression (HIV RNA < 50 copies/mL) at 12 Months after Initiating or Switching to B/F/TAF | 12 Months

SECONDARY OUTCOMES:
Percentage of Participants with HIV-1 RNA Suppression (HIV RNA < 50 copies/mL) at 3 Months After Initiating or Switching to B/F/TAF | 3 Months
Proportion of Participants with HIV-1 RNA Suppression (HIV RNA < 50 copies/mL) at 6 Months After Initiating or Switching to B/F/TAF | 6 Months
Percentage of Participants with HIV-1 RNA Suppression (HIV RNA < 50 copies/mL) at 24 Months After Initiating or Switching to B/F/TAF | 24 Months
Change in CD4 Cell Count at 3 Months After Initiating or Switching to B/F/TAF | 3 Months
Change in CD4 Cell Count at 6 Months After Initiating or Switching to B/F/TAF | 6 Months
Change in CD4 Cell Count at 12 Months After Initiating or Switching to B/F/TAF | 12 Months
Change in CD4 Cell Count at 24 Months After Initiating or Switching to B/F/TAF | 24 Months
CD4/CD8 Ratio at 3 Months After Initiating or Switching to B/F/TAF | 3 Months
CD4/CD8 Ratio at 6 Months After Initiating or Switching to B/F/TAF | 6 Months
CD4/CD8 Ratio at 12 Months After Initiating or Switching to B/F/TAF | 12 Months
CD4/CD8 Ratio at 24 Months After Initiating or Switching to B/F/TAF | 24 Months
Percentage of Participants Experiencing Adverse Events and Serious Adverse Events | 24 Months

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (5):
- Israel (5):
  - Rambam Medical Center, Haifa
  - Hadassah Medical Center, Jerusalem
  - Kaplan Medical Center, Rehovot
  - Tel Aviv Souraski Medical Center, Tel Aviv
  - Sheba Medical Center, Tel Litwinsky

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Antinori A, Yokomaku Y, Elinav H, Pullukcu H, de Wet J, Antela A, Lu PL, Sabranski M, Kim YS, Bonnet F, den Hollander J, Jackson A, Choy CY, Cai W, Zhang F, Thorpe D, Marongiu A, Harrison R, Jarrett J, Boffito M. Quality of Life and Treatment Satisfaction in People with HIV Switching to Bictegravir/Emtricitabine/Tenofovir Alafenamide: Pooled Analysis from Observational Cohort Studies. Infect Dis Ther. 2026 Jan;15(1):217-244. doi: 10.1007/s40121-025-01252-w. Epub 2025 Nov 24. PMID 41284214